CLINICAL TRIAL: NCT04826601
Title: The Physical and Psychologic Effects of Aromatherapy in Cancer Patients During Chemotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Show Chwan Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chun-Yi Lin, Dr., Show Chwan Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SRD-109037
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Pain; Heart Rate Variability; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Oils, Volatile

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental)
  Interventions: Other: essential oils

INTERVENTIONS:
Other: essential oils — A total of 40 cancer patients receiving chemotherapy will be recruited as participants in this study. Blood orange and rosewood will be chosen as the essential oils for aromatherapy in this study. Essential oils will be applied to all participants by inhalation for 30 minutes.

SUMMARY:
Background: Stress is the critical method for survive of reacting to a condition including a threat, challenge or physical and psychological challenge. Stress either physiological or biological is an organism's response to a stressor such as an environmental condition. Stimuli that alter an organism's environment are responded to by multiple systems in the body. The hypothalamic-pituitary-adrenal (HPA) axis and autonomic nervous system are major systems which the body reacts to the stress. It has been reported that cancer patients receiving chemotherapy perceived a lot of stress. It has been believed and well known that stress-related illness is one of the reasons contributing to the increase in long-term sick leave during the last decade in many countries.

Purpose: The aims of this study are to evaluate the effects of aromatherapy on cancer patient receiving chemotherapy: 1) for physical effects by meridian electrical conductance, heart rate variability (HRV), vital sign, visual analogue scale (VAS) for pain; 2) for psychologic effects by State-Trait Anxiety Inventory (STAI).

Materials and methods: This is a prospective, pre post comparison study. A total of 40 cancer patients receiving chemotherapy will be recruited as participants in this study. The characteristics data will be collected in all participants. Blood orange and rosewood will be chosen as the essential oils for aromatherapy in this study. Essential oils will be applied to all participants by inhalation for 30 minutes. Meridian electrical conductance, HRV, vital sign, VAS for pain, and STAI were evaluated and compared before and after aromatherapy.

Expected outcomes: It is expected to understand more about the effects of aromatherapy on the meridian system, HRV and emotional status by undertaking 30 minutes session aromatherapy intervention for cancer patients receiving chemotherapy. The results may suggest aromatherapy as one of the affiliated programs of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* cancer patients in chemotherapy
* Subjects who are aged from 20 to 70 years-old

Exclusion Criteria:

* Subjects who are unable to read and sign the consent form
* diagnosed with a major illness (such as acute myocardial infarction, stroke, paralysis, and major organ transplantation)
* being pregnant

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-05-12 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
pain score | immediately after aromatherapy
  Visual analogue scale for pain. Scores are recorded between 0 for "no pain" and 10 for "worst pain". A higher score indicates greater pain intensity.

SECONDARY OUTCOMES:
Anxiety | immediately after aromatherapy
  State-Trait Anxiety Inventory (STAI)

CONTACTS AND LOCATIONS:
Locations (1):
- Show Chwan Memorial Hospital, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farahani MA, Afsargharehbagh R, Marandi F, Moradi M, Hashemi SM, Moghadam MP, Balouchi A. Effect of aromatherapy on cancer complications: A systematic review. Complement Ther Med. 2019 Dec;47:102169. doi: 10.1016/j.ctim.2019.08.003. Epub 2019 Aug 5. PMID 31779991
- [Background] POKORNY AD, MOORE FJ. Neuroses and compensation: chronic psychiatric disorders following injury or stress in compensable situations. I. Review of the literature. AMA Arch Ind Hyg Occup Med. 1953 Dec;8(6):547-63. No abstract available. PMID 13103829
- [Background] MIKUTA JJ, PAYNE FL. Stress urinary incontinence in the female; a review of the modern approach to this problem. Am J Med Sci. 1953 Dec;226(6):674-87. doi: 10.1097/00000441-195312000-00010. No abstract available. PMID 13104420
- [Background] VEILLEUX R. THE STRESS CONCEPT AS WE SEE IT TODAY. Adv Vet Sci. 1963;8:189-213. No abstract available. PMID 14272336
- [Background] RAJUSZ E. NEUROENDOCRINE RELATIONSHIPS. Prog Neurol Psychiatry. 1963;18:306-47. No abstract available. PMID 14146314